CLINICAL TRIAL: NCT01142167
Title: A Study to Assess the Success Rate of Ultra-thin Colonoscopy Versus Conventional Colonoscopy for the First or Rescue Colonoscopy for Unsuccessful Procedures (UTC Study).
Brief Title: A Comparison of an Ultra-thin and Standard Colonoscope in Achieving Caecal Intubation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: UTC Study
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: First Colonoscopy Examination
Keywords: Ultra-thin colonoscope

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Colonoscopy (Active Comparator): Colonoscopy with standard instrument
  Interventions: Procedure: Standard Colonoscopy
- Ultra-thin colonoscopy (Experimental): New prototype scope
  Interventions: Procedure: Ultra-thin colonoscopy

INTERVENTIONS:
Procedure: Standard Colonoscopy — Standard colonoscopy will be used during colonoscopy
  Arms: Standard Colonoscopy
Procedure: Ultra-thin colonoscopy — Ultra-thin colonoscope will be used during colonoscopy
  Arms: Ultra-thin colonoscopy

SUMMARY:
The aim of the study is to study the caecal intubation rate of a prototype ultra-thin colonoscope compared to a standard colonoscope and to study usefulness of this new colonoscope as a rescue instrument for failed initial colonoscopy with a standard colonoscope and to study the patient satisfaction scores using a validated endoscopy GHAA-9 for a new prototype colonoscope as compared to a standard colonoscope.

DETAILED DESCRIPTION:
Colonoscopy is a common endoscopic procedure, widely used for the investigation of lower gastrointestinal tract diseases manifesting as altered bowel habit, per rectal bleeding and abdominal pain. It is used to diagnose colonic polyps, colorectal cancer and inflammatory bowel disease to name a few examples.

Colorectal cancer screening has been shown to decrease colorectal cancer. Despite this the uptake by the general population is suboptimal.

A new prototype colonoscope from Olympus with an additional distal bending section was designed. The investigators hypothesize that its performance characteristics will be similar to a standard colonoscope with patient tolerability.

This randomised control trial aims to invite patients attending their first outpatient colonoscopy and who are able to provide informed consent.(so they have had no prior experience) to assess the completion rate, patient and endoscopist satisfaction.

Patients with prior colorectal surgery or previous colonoscopy were excluded.

ELIGIBILITY:
Inclusion Criteria:

* First outpatient colonoscopy
* Able to provide informed consent

Exclusion Criteria:

* Unable to provide consent
* Prior colon surgery (except appendectomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1121 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Successful Caecal intubation | 12 weeks
  Success of Caecal intubation for the ultra-thin colonoscope vs standard colonoscope

SECONDARY OUTCOMES:
Caecal intubation time | 12 weeks
  Caecal intubation time Ultra-thin colonsocope vs standard colonoscope
Patient Satisfaction and Pain score | 12 weeks
  Patient tolerability Ultra-thin vs standard colonoscope
Endoscopist satisfaction | 12 weeks
  Ease of use prototype scope vs standard colonoscope

CONTACTS AND LOCATIONS:
Overall Officials: James Y Lau, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Endoscopy Center, Prince of Wales Hospital, Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Luo DJ, Hui AJ, Yan KK, Ng SC, Wong VW, Chan FK, Cheong JP, Lam PP, Tse YK, Lau JY. A randomized comparison of ultrathin and standard colonoscope in cecal intubation rate and patient tolerance. Gastrointest Endosc. 2012 Mar;75(3):484-90. doi: 10.1016/j.gie.2011.07.032. Epub 2011 Oct 1. PMID 21963069